CLINICAL TRIAL: NCT05972174
Title: Phase 1/2, Randomized, Observer-Blind, Parallel, Dose-Ranging Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1018 Pandemic Influenza Candidate Vaccines in Healthy Adults ≥18 Years of Age
Brief Title: A Study of mRNA-1018 Pandemic Influenza Candidate Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1018-P101
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Influenza
Keywords: Influenza vaccine; Moderna; mRNA-1018; Virus Diseases; Vaccines; Pandemic influenza
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Part A Group 1 Vaccine: mRNA-1018 for H5N8 Dose Level 1 (Experimental): Participants will receive mRNA-1018 for H5N8 at dose level 1 by intramuscular (IM) injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H5N8
- Part A Group 1 Vaccine: mRNA-1018 for H5N8 Dose Level 2 (Experimental): Participants will receive mRNA-1018 for H5N8 at dose level 2 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H5N8
- Part A Group 1 Vaccine: mRNA-1018 for H5N8 Dose Level 3 (Experimental): Participants will receive mRNA-1018 for H5N8 at dose level 3 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H5N8
- Part A Group 1 Vaccine: mRNA-1018 for H5 Only Dose Level 1 (Experimental): Participants will receive mRNA-1018 for H5 only at dose level 1 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H5 Only
- Part A Group 1 Vaccine: mRNA-1018 for H5 Only Dose Level 2 (Experimental): Participants will receive mRNA-1018 for H5 only at dose level 2 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H5 Only
- Part A Group 1 Vaccine: mRNA-1018 for H5 Only Dose Level 3 (Experimental): Participants will receive mRNA-1018 for H5 only at dose level 3 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H5 Only
- Part A Group 2 Vaccine: mRNA-1018 for H7N9 Dose Level 1 (Experimental): Participants will receive mRNA-1018 for H7N9 at dose level 1 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H7N9
- Part A Group 2 Vaccine: mRNA-1018 for H7N9 Dose Level 2 (Experimental): Participants will receive mRNA-1018 for H7N9 at dose level 2 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H7N9
- Part A Group 2 Vaccine: mRNA-1018 for H7N9 Dose Level 3 (Experimental): Participants will receive mRNA-1018 for H7N9 at dose level 3 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H7N9
- Part A Group 2 Vaccine: mRNA-1018 for H7 Only Dose Level 1 (Experimental): Participants will receive mRNA-1018 for H7 only at dose level 1 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H7 Only
- Part A Group 2 Vaccine: mRNA-1018 for H7 Only Dose Level 2 (Experimental): Participants will receive mRNA-1018 for H7 only at dose level 2 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H7 Only
- Part A Group 2 Vaccine: mRNA-1018 for H7 Only Dose Level 3 (Experimental): Participants will receive mRNA-1018 for H7 only at dose level 3 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H7 Only
- Part B Group 1 Vaccine: mRNA-1018 for H5 Only-CG Dose Level 1 (Experimental): Participants will receive mRNA-1018 for H5 Only-CG at dose level 1 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H5 Only-CG
- Part B Group 1 Vaccine: mRNA-1018 for H5 Only-CG Dose Level 2 (Experimental): Participants will receive mRNA-1018 for H5 Only-CG at dose level 2 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H5 Only-CG
- Part B Group 1 Vaccine: mRNA-1018 for H5 Only-CG Dose Level 3 (Experimental): Participants will receive mRNA-1018 for H5 Only-CG at dose level 3 by IM injection on Day 1 and Day 22.
  Interventions: Biological: mRNA-1018 for H5 Only-CG

INTERVENTIONS:
Biological: mRNA-1018 for H5N8 — Sterile liquid for injection
  Arms: Part A Group 1 Vaccine: mRNA-1018 for H5N8 Dose Level 1; Part A Group 1 Vaccine: mRNA-1018 for H5N8 Dose Level 2; Part A Group 1 Vaccine: mRNA-1018 for H5N8 Dose Level 3
Biological: mRNA-1018 for H7N9 — Sterile liquid for injection
  Arms: Part A Group 2 Vaccine: mRNA-1018 for H7N9 Dose Level 1; Part A Group 2 Vaccine: mRNA-1018 for H7N9 Dose Level 2; Part A Group 2 Vaccine: mRNA-1018 for H7N9 Dose Level 3
Biological: mRNA-1018 for H5 Only — Sterile liquid for injection
  Arms: Part A Group 1 Vaccine: mRNA-1018 for H5 Only Dose Level 1; Part A Group 1 Vaccine: mRNA-1018 for H5 Only Dose Level 2; Part A Group 1 Vaccine: mRNA-1018 for H5 Only Dose Level 3
Biological: mRNA-1018 for H7 Only — Sterile liquid for injection
  Arms: Part A Group 2 Vaccine: mRNA-1018 for H7 Only Dose Level 1; Part A Group 2 Vaccine: mRNA-1018 for H7 Only Dose Level 2; Part A Group 2 Vaccine: mRNA-1018 for H7 Only Dose Level 3
Biological: mRNA-1018 for H5 Only-CG — Sterile liquid for injection
  Arms: Part B Group 1 Vaccine: mRNA-1018 for H5 Only-CG Dose Level 1; Part B Group 1 Vaccine: mRNA-1018 for H5 Only-CG Dose Level 2; Part B Group 1 Vaccine: mRNA-1018 for H5 Only-CG Dose Level 3

SUMMARY:
The purpose of this Phase 1/2 study is to generate sufficient safety and immunogenicity data of mRNA-1018 pandemic influenza candidate vaccines in healthy adults ≥18 years of age to enable the initiation of a large Phase 3 trial with one selected vaccine candidate. The study will be conducted in 2 Parts (Part A and Part B) that will enroll and run concurrently. Part A of the study will evaluate 4 vaccine candidates (H5N8, H7N9, H5 only, and H7 only). Part B of the study will evaluate a single vaccine candidate (H5 only-CG).

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and results of electrocardiogram testing.
* Body mass index of 18 kilograms (kg)/square meter (m^2) to 39 kg/m^2 (inclusive) at the Screening visit.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception, and not currently breastfeeding.

Key Exclusion Criteria:

* Participant is acutely ill or febrile (body temperature ≥ 38.0 degrees Celsius [°C]/100.4 degrees Fahrenheit [°F]) 72 hours prior to or at the Screening Visit or Day 1.
* History of a diagnosis or condition that, in the judgment of the Investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures.
* Any medical, psychiatric, or occupational condition, including reported history of substance abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Participant has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 180 days prior to Screening Visit (for corticosteroids ≥10 milligrams [mg]/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
* Participant has received any vaccine authorized or approved by local health agency including mRNA vaccine ≤28 days prior to study intervention (Day 1) or plans to receive a vaccine authorized or approved by local health agency within 28 days before or after the study intervention.
* Participant has participated in an interventional clinical study within 28 days prior to the Screening visit based on the medical history interview or plans to do so while participating in this study.

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1504 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to Day 29 (7 days after each injection)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 43 (21 days after each injection)
Number of Participants with AEs Leading to Discontinuation From Study | Day 1 to Day 205 (end of study [EoS])
Number of Participants with Medically-Attended AEs (MAAEs) | Day 1 to Day 205 (EoS)
Number of Participants with Serious Adverse Events (SAEs) | Day 1 to Day 205 (EoS)
Number of Participants with Adverse Events of Special Interest (AESIs) | Day 1 to Day 205 (EoS)

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of Anti-Hemagglutinin (HA) Antibodies at Days 22, 29, and 43, as Measured by Hemagglutination Inhibition (HAI) Assay | Days 22, 29, and 43
Geometric Mean Fold Rise (GMFR) of Anti-HA Antibodies From Baseline to Days 22, 29, and 43, as Measured by HAI Assay | Baseline (Day 1), Days 22, 29, and 43
Number of Participants With Seroconversion at Days 22, 29, and 43, as Measured by HAI Assay | Baseline (Day 1) to Days 22, 29, and 43
  Seroconversion is defined as a Day 22, 29, or 43 titer ≥1:40 if baseline is <1:10 or a 4-fold or greater rise if baseline is ≥1:10 in anti-HA antibodies measured by HAI assay.
Number of Participants With HAI Titer ≥ 1:40 at Days 22, 29, and 43 | Days 22, 29, and 43
GMT of Anti-Neuraminidase (NA) Antibodies at Days 22, 29, and 43, as Measured by Neuraminidase Inhibition (NAI) Assay | Days 22, 29, and 43
GMFR of Anti-NA Antibodies From Baseline to Days 22, 29, and 43, as Measured by NAI Assay | Baseline (Day 1), Days 22, 29, and 43
Number of Participants with a Change in the Days 22, 29, and 43 NAI Titer of at Least 2-/3-/4-Fold Rise | Baseline (Day 1) to Days 22, 29, and 43
  Number of participants with a change in the Days 22, 29, or 43 NAI titer of at least 2-/3-/4-fold rise, defined as ≥2-/3-/4-fold of the lower level of quantitation (LLOQ) if the Day 1 titer is <LLOQ; or ≥2-/3-/4-fold of the Day 1 titer if the Day 1 titer is ≥LLOQ.

CONTACTS AND LOCATIONS:
Locations (27):
- United States (9):
  - CenExel RCA, Hollywood, Florida
  - Velocity Clinical Research, Savannah, Georgia
  - Johnson County Clin-Trials, Lenexa, Kansas
  - DM Clinical Research, Southfield, Michigan
  - Velocity Clinical Research, Lincoln, Nebraska
  - Velocity Clinical Research Providence, East Greenwich, Rhode Island
  - DM Clinical Research, Sugar Land, Texas
  - DM Clinical Research, Tomball, Texas
  - J. Lewis Research, Inc/Jordan River Family Medicine, South Jordan, Utah
- United Kingdom (18):
  - Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Southampton General Hospital, Southampton, England
  - University Hospitals Birmingham, Birmingham, London
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford, London
  - University Hospitals, Bristol, London
  - Cardiff and Vale University, Cardiff, London
  - Northern Care Alliance, Salford, London
  - Royal Cornwall Hospital, Truro, London
  - North Wales Clinical Research Centre, Wrexham, London
  - Quadram Institute NNUH CRF, Norwich, Norfolk
  - Lakeside Healthcare Research Unit, Corby, Northamptonshire
  - Western Hospital Edinburgh, Edinburgh
  - Royal Free Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust - St Thomas' Hospital, London
  - Chelsea and Westminster Hospital, London
  - St Georges Vaccine Institute Cranmer Terrace, London
  - University College London Hospitals NHS Foundation Trust, London
  - Velocity Clinical Research, North Finchley